CLINICAL TRIAL: NCT04909099
Title: Cross-cultural Adaptation and Psychometric Properties of the Arabic Version of the Exercise Adherence Rating Scale
Brief Title: Arabic Version of the EARS Questionnaire
Acronym: EARS-Ar
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Prince Sultan Military College of Health Sciences (Other)
Collaborators: King Fahd Military Medical Complex (Unknown)
Responsible Party: Principal Investigator, Ahmed Farrag, Assisstant Professor, Prince Sultan Military College of Health Sciences
Other Study IDs: IRB-2020-PT-039
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Knee Osteoarthritis; Low Back Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Knee Ostearthritis/ Low Bakc Pain: Patients referred for physical therapy rehabilitation
  Interventions: Other: Standard treatment

INTERVENTIONS:
Other: Standard treatment — Participants shall fill the EARS-Ar questionnaire three times within one month in addition to other questionnaires including the Roland Morris Disability Questionnaire (RMDQ) for low back pain (LBP) patients, and the Knee injury and Osteoarthritis Outcome Score (KOOS) for knee OA patients, in addition to the Fear-Avoidance Beliefs Questionnaire (FABQ), the Numeric Pain Rating Scale (NPRS), and the Global Rating of Change Scale (GRoC).
  The first time will be one week after enrolling in the study and receiving the prescribed home exercise program. the second time will be 3-6 days later to test the reliability of the EARS-Ar. After another week, participants will refill the EARS-Ar and the GRoC to test responsiveness.

SUMMARY:
A study to translate and cross-culturally adapt the Exercise Adherence Rating Scale (EARS) into the Arabic language, and assess its psychometric properties.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain patients: aged 18 years or older, experienced non-specific CLBP of 3 months or longer, pain localized to the lumbar region.
* Knee OA patients: eligible participants must meet the knee OA diagnostic criteria according to the American College of Rheumatology (ACR).

Exclusion Criteria:

* degenerative systemic diseases
* neurological symptoms
* lumbar stenosis
* spondylolisthesis
* history of spinal or knee surgeries
* pregnancy
* rheumatoid arthritis
* serious pathological conditions (inflammatory arthritis and malignancy)
* individuals who cannot read and understand documents written in the Arabic language.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential participants will be recruited from patients with chronic low back pain (CLBP) or knee osteoarthritis referred to the outpatient physical therapy services of the local medical facilities.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Floor and ceiling effect | 1 day
  It will be considered present if more than 15% of the sample score the lowest or highest possible total score, respectively
Content Validity | 1 day
  Assessed using the Content Validity Index (CVI) with an acceptable value of at least 0.8.
Construct Validity | 1 day
  Assessed by calculating the Spearman's correlation coefficient (ρ) between the Exercise Adherence Rating Scale-Arabic version (EARS-Ar) score and the Fear Avoidance Belief Questionnaire (FABQ), the Numeric Pain Rating Scale (NPRS), the Roland-Morris Disability Questionnaire (RMDQ), and the Knee Injury and osteoarthritis Outcome Score (KOOS) measurement tools. The coefficient is classified as follows: ρ = 0.3-0.7 moderate correlation, and >0.7 strong correlation.
Internal Consistency | 3-7 days
  Assessed by calculating the Cronbach's alpha (α) and the corrected item-total correlation. A Cronbach's α value of ≥0.7, and a corrected item-total correlation, measured using the Pearson correlation coefficient, of ≥0.3 will be considered acceptable.
Test-retest Reliability | 3-7 days
  Assessed by calculating the intraclass correlation coefficient (ICC) between the EARS-Ar scores of the first two test sessions. An ICC value of >0.8 and 0.6-0.8 will be considered as excellent and good correlation, respectively.

SECONDARY OUTCOMES:
Responsiveness | 3 weeks
  Participating patients will be categorized according to their reported Global Rating of Change (GRoC) scores (external anchor) to either improved (GRoC≥3) or stable group (GRoC<3 to >-3) and a between-group comparison will be performed using an unpaired t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Farrag, PhD, Principal Investigator — Cairo University
Locations (1):
- King Fahd Military Medical Complex, Dhahran, Eastern Province, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Background] Meade LB, Bearne LM, Godfrey EL. Comprehension and face validity of the Exercise Adherence Rating Scale in patients with persistent musculoskeletal pain. Musculoskeletal Care. 2018 Sep;16(3):409-412. doi: 10.1002/msc.1240. Epub 2018 Mar 25. No abstract available. PMID 29575381
- [Background] Terwee CB, Bot SD, de Boer MR, van der Windt DA, Knol DL, Dekker J, Bouter LM, de Vet HC. Quality criteria were proposed for measurement properties of health status questionnaires. J Clin Epidemiol. 2007 Jan;60(1):34-42. doi: 10.1016/j.jclinepi.2006.03.012. Epub 2006 Aug 24. PMID 17161752
- [Background] Newman-Beinart NA, Norton S, Dowling D, Gavriloff D, Vari C, Weinman JA, Godfrey EL. The development and initial psychometric evaluation of a measure assessing adherence to prescribed exercise: the Exercise Adherence Rating Scale (EARS). Physiotherapy. 2017 Jun;103(2):180-185. doi: 10.1016/j.physio.2016.11.001. Epub 2016 Nov 9. PMID 27913064
- [Background] de Lira MR, de Oliveira AS, Franca RA, Pereira AC, Godfrey EL, Chaves TC. The Brazilian Portuguese version of the Exercise Adherence Rating Scale (EARS-Br) showed acceptable reliability, validity and responsiveness in chronic low back pain. BMC Musculoskelet Disord. 2020 May 12;21(1):294. doi: 10.1186/s12891-020-03308-z. PMID 32398068